CLINICAL TRIAL: NCT01933646
Title: Burden of Invasive Group B Streptococcal (GBS) Disease in Young Infants in China: Incidence, Case Fatality Rate and Serotype Distribution
Brief Title: Burden of Invasive Group B Streptococcal (GBS) Disease in Young Infants in China
Status: Completed | Type: Observational
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: V98_23OB
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Invasive Group B Streptococcal Disease
Keywords: Group B streptococcus; Incidence; Case fatality rate; Serotype distribution

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1

SUMMARY:
Evaluate the burden of invasive group B streptococcal (GBS) disease in young infants (up to 90 days of age) in China, in terms of incidence, case fatality rate and serotype distribution

ELIGIBILITY:
Inclusion Criteria:

1. Positive culture for GBS from one or more of the following normally sterile sites: blood, cerebrospinal fluid (CSF), pleural fluid, peritoneal fluid, pericardial fluid, surgical aspirate, bone, joint fluid, suprapubic bladder aspiration or internal body site (e.g., lymph node, brain).
2. ≤90 days old at the time of GBS confirmation.
3. Voluntary written informed consent provided.

Exclusion Criteria:

* None.

Max Age: 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants (up to and including 90 days of age) born in or treated in a study hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incidence of group B streptococcal (GBS) disease | From birth to 90 days of age
Case Fatality Rate of GBS disease | From birth to 90 days of age
GBS serotype distribution | From birth to 90 days of age

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (3):
- China (3):
  - Site 12, Changsha
  - Site 13, Guangzhou
  - Site 14, Guangzhou

REFERENCES:
- [Background] Heath PT, Schuchat A. Perinatal group B streptococcal disease. Best Pract Res Clin Obstet Gynaecol. 2007 Jun;21(3):411-24. doi: 10.1016/j.bpobgyn.2007.01.003. Epub 2007 Mar 2. PMID 17336588